CLINICAL TRIAL: NCT06069128
Title: A Single Center, Open Label, Pilot Study to Evaluate the Usability of the Neuro-trigger Artificial Eye Blinking Stimulation Device in Patients With Paralysis of the Facial Nerve.
Brief Title: Evaluate the Usability of the Neuro-trigger Artificial Eye Blinking Stimulation Device in Patients With Paralysis of the Facial Nerve.
Acronym: paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurotrigger Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0100
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Paralysis; Paralysis; Eye; Paralysis; Bell
MeSH Terms: conditions — Paralysis; Bell Palsy

STUDY DESIGN:
Intervention Model Description: This is a single-center, open label clinical study. Up to 11 subjects will be enrolled to use the Neuro-trigger device for blinking stimulation for a duration of 14 days.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neurotrigger device treatment arm (Experimental): treatment with Neuro-trigger device for blinking stimulation for a duration of 14 days
  Interventions: Device: Neurotrigger Basic. eye blinking stimulator

INTERVENTIONS:
Device: Neurotrigger Basic. eye blinking stimulator — NeuroTrigger Basic is intended to stimulate healthy muscles in order to improve or facilitate muscle performance for maintaining/increasing muscle range of motion and for the prevention or retardation of disuse atrophy.
  Other Names: NTB-KT-0003

SUMMARY:
This is a single-center, open-label clinical study. Up to 11 subjects will be enrolled to use the Neuro-trigger device for blinking stimulation for a duration of 14 days.

DETAILED DESCRIPTION:
Facial paralysis is a well-known and severe condition. The paralysis can be permanent or temporary, depending on the cause and on the severity. It usually affects only one side of the patient's face, and so it makes the affected side of the face look like it is drooping.

The two facial nerves control each the muscles on one side of the face. A damaged facial nerve distal to the impaired area is dead and is unable to carry messages from the brain to the facial respective muscles either completely or partially, depending on the level of damage. This leads to muscle weakness, twitching or paralysis. In addition, damage to the nerve can cause the eyelid to drop, and the angle of the patient's mouth can also be twisted, usually towards down. In some cases of bell's Palsy, the nerve is capable to regenerate into the tunnel where it run before, and some studies have shown that stimulation may facilitate the growth toward the desired direction.

Under normal circumstances, the human eye blinks every 2-10 seconds. With every blink the eyelid spreads moisture over the cornea. With facial paralysis the ability to blink may be impaired or absent all together.The dry eye syndrome gets exacerbated since damage to the facial nerve also impairs the signal to the tear gland to generate tears, which mean that the production and secretion of tears in the affected eye is impaired.

With no effective treatment so far, and as paralysis persists, the severity of secondary damage to the eye increases including irritation of the eye (conjunctivitis), ulceration of the cornea, and it might cause severe disability and even blindness.

All the treatment options currently offered in the cases described above are partial and insufficient, and are aimed at alleviating symptoms and providing relief only.

The current treatment options are:

1. Application of eye drops (artificial tears), gel and\or ointment
2. Tarsorrhaphy is the surgical fusion of the upper and lower eyelid margins.
3. Eyelid gold weight insertion.
4. A punctual plug.

Most of the existing treatment options deal with the symptoms of the dry eye syndrome, such as blurred vision, while the solution proposed by us is designed to address the original cause of the problem - the loss of eye muscle blinking due to loss of nerve stimulus due to the injury of the facial nerve.

The Neurotrigger device offers a comprehensive treatment system mainly designed for cases of functional impairment of the eye due to facial paralysis.

People with facial nerve paralysis cannot blink and cannot close the affected eye, day or night. As a result, the patients suffer from short and long-term consequences, including pain, discomfort, dry eye syndrome, and possible graduate impairment of vision.

Therefore, we suggest a novel daytime stimulating device based on an electrical stimulation of the facial nerve designed to restore blinking. This device is estimated to advance/improve/create a breakthrough in the current available treatment for rehabilitation of the affected eye in cases of facial nerve paralysis.

We recommend using this novel daytime system in combination with a specific solution for nighttime, designed to mechanically maintain the eye closed at night.

The day and night component of the solution have each separately its specific merits yet combining both solutions, creates a comprehensive treatment that may bring clear improvement for the patient.

The Neurotrigger device aims to restore eye blinking during the day based on electrical stimulation that is carried by the underlying injured nerve to activate the respective muscle unit and renew eye blinking and tear release.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects above 18 years of age
* Subject whom able to provide a written informed consent.
* Subjects who are willing to provide medical and demographic records of their facial paralysis, the consequences of the paralysis and general medical history.
* Patients who answer the full definition of continuous existing unilateral facial paralysis.
* Patients who comply with the definition of unilateral facial paralysis up to 12 months from the first diagnosis.
* Enrolment will depend on the subject's willingness and capability to perform the daily treatment with the use of the Neuro-trigger simulator (including operating the device and electrode placement ) for a duration of 2 weeks.

Exclusion Criteria:

* Patients with chronic facial paralysis and secondary established damage to the eye occurring prior to enrollment, who did not undergo facial reanimation surgery.
* Patients with psychiatric, addictive, or any other disorder that compromises ability to give genuine informed consent for participation in this study.
* Patients suffering from any skin condition that will prevent effective attachment of the electrodes, including but not limited to allergy to any of the components of the skin electrode
* Woman who is pregnant (positive pregnancy test)
* Woman who is nursing
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Patients who underwent an operation for facial reanimation at least one year prior to enrollment
* Patients whom are currently participating in other clinical study
* High probability of orbicularis oculi atrophy or damage (i.e. long-standing facial paralysis or cases
* History of ablative surgery where the musculature has been sacrificed)
* History of prior facial reanimation procedures
* History of diabetic neuropathy, unstable cardiovascular disease, neurologic disease causing severe
* cognitive or motor impairment, severe immunological deficiency, and malignant diseases that are not in remission
* Signs of corneal infection or severe ocular surface inflammation
* Cardiac demand pacemaker, implanted defibrillator or other implanted electronic device

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the Neuro-trigger device usability in the treatment of unilateral facial paralysis subjects. | 14 days treatment
  Examining the optimal location of placement for the Neuro- trigger's electrodes.
  * Establishing the level of pain generated if any, during device implementation and stimulation.
  * Exploring the personal adjustment process of the precise pattern of stimulation (strength, intensity, other features) to achieve eye blinking for different patients

SECONDARY OUTCOMES:
The secondary study objective is to evaluate the safety and effectiveness of the BlinkER in achieving eyelid closure during the study visits with facial nerve palsy. | 14 days treatment
  * The number reported related of serious adverse events occurring throughout the study participation duration.
  * The number of reported related Adverse events occurring throughout the study participation duration.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Keidar, Dr, Principal Investigator — Tel Aviv sourasky medical center ichilov
Locations (1):
- Tel Aviv Sourasky Medical Center (Ichilov), Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided